CLINICAL TRIAL: NCT07146672
Title: Exploratory Study of Super DC Cell Injection in Preventing Recurrence After Radical Surgery for Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BZT003-A-03
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor Cancer
Keywords: Vaccines; Immunologic Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): A single dose of 1×10^7 cells, with a dosing interval of 1 week or 2 weeks during the induction period.
  Interventions: Biological: Super DC Vaccine
- Group 2 (Experimental): A single dose of 2×10^7 cells, with a dosing interval of 1 week or 2 weeks during the induction period.
  Interventions: Biological: Super DC Vaccine

INTERVENTIONS:
Biological: Super DC Vaccine — Super DC Cell Injection

SUMMARY:
The study is a controlled, open-label exploratory clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, weight ≥ 40kg; No gender limit；
* Subjects with malignant solid tumors diagnosed by histology or cytology and undergoing radical resection surger；
* At the beginning of the study (after surgery), there were no lesions, no local recurrence or distant metastasis on the imaging, and no brain metastasis (images within one month before enrollment can be used for screening)；
* Subjects in the safety verification stage need to provide immunohistochemical test results with positive expression of Survivin or P53 or MUC1;
* ECOG score 0-1 points;
* There are sufficient venous channels and no contraindications for peripheral blood mononuclear cell collection surgery;
* Organs and bone marrow function well:
* a:Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50% evaluated by echocardiography within one month of enrollment; The electrocardiogram is basically normal;
* b:Platelets ≥ 90 × 10 ^ 9/L;
* c:Hemoglobin ≥ 90g/L (no blood transfusion or erythropoietin dependence within 7 days);
* d:Total bilirubin ≤ 2 times the upper limit of normal value;
* e:Serum creatinine ≤ 1.5 times the upper limit of normal value;
* f:Transaminases (AST, ALT) ≤ 2.5 times the upper limit of normal value (if liver cancer is 5 times the upper limit of normal value);
* g:International standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times the upper limit of normal value;
* Able to understand trial requirements and matters, willing to participate in clinical research according to trial requirements

Exclusion Criteria:

* Positive for HIV antibodies or syphilis antibodies; positive for hepatitis B surface antigen, and positive for hepatitis B core antibody or e antibody with viral DNA copy number above the detection limit or ≥1000 copies/ml; or hepatitis C virus RNA copy number above the detection limit.
* Any uncontrollable active infection, coagulation disorder, or any other major disease;
* Pregnant or lactating women;
* Suffering from active neuroautoimmune or inflammatory diseases, such as any of the following: inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, multiple sclerosis, Sjogren's syndrome, etc., and receiving relevant treatment; Subjects who are still using immunosuppressants for organ transplantation; Or subjects who have been using immunosuppressive drugs such as glucocorticoids for a long time cannot stop at least 4 weeks before enrollment; Severe allergic constitution;
* Subjects with existing abnormalities in the central nervous system, such as seizures, cerebral vascular ischemia/bleeding, dementia, cerebellar diseases, or any autoimmune diseases associated with central nervous system involvement;
* Major cardiovascular diseases with clinical significance include:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Within 28 days after the first injection
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mengchao Tumor Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No